CLINICAL TRIAL: NCT05098392
Title: Effects of Sibling-Mediated Intervention on Early Literacy and Social Reciprocity for Children With Autism
Brief Title: Sibling-Mediated Intervention on Literacy and Reciprocity for Children With Autism
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in recruiting required participants.
Sponsor: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00014411
Record Dates: First submitted 2021-10-13; First posted 2021-10-28 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Children in the US and China will be randomized into the two groups at each location.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will not be informed of the group status of the children.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual/Sibling interaction (No Intervention): Children with autism will spend time with their typically developing siblings for 20-30 mins at least three times a week
- Sibling-mediated intervention (Experimental): Children with autism will receive explicit instruction from their typically developing siblings
  Interventions: Behavioral: Sibling-mediated intervention

INTERVENTIONS:
Behavioral: Sibling-mediated intervention — Typically developing siblings will be trained to use an explicit instruction strategy (model-lead-test) and a checklist to self-monitor their teaching when working with their siblings with ASD on reading and social skills.
  Arms: Sibling-mediated intervention

SUMMARY:
Given the increasing prevalence of autism spectrum disorder (ASD), estimated to be 1 in 68 in the United States alone, ASD has become one of the fastest-growing pediatric concerns. The deficits of children with ASD range across social communication and academic skills. One of the effective interventions that have been used commonly for ASD is the model-lead-test, which includes modeling, prompting children to practice target skills together, and providing children with affirmative feedback or error correction. Previous research has demonstrated that the model-lead-test is successful in teaching different skills for individuals with ASD, including functional, social, and academic skills. The vast majority of the studies had researchers, therapists, or teachers implement the intervention. However, there is clear empirical support and implications for interventions mediated by more familiar persons, such as parents and siblings, which may lead to better effects, maintenance, and generalization due to more practice opportunities in the natural environments. Research has supported the effectiveness of using parents or peers as agents to deliver interventions for individuals with ASD, whereas fewer studies explored the use of siblings to deliver or mediate intervention. As typically developing siblings are an essential part of the daily life of children with ASD, it makes logical extensions to have siblings as mediators to deliver interventions.

In the initial findings, the investigators found the typically developing siblings can accurately implement the model-lead-test procedure that improved various skills of their siblings with ASD. This project will extend these findings by examining the efficacy of the sibling-implemented intervention on early literacy (reading) and social reciprocity (conversation and play) of children with ASD as well as the sibling relationship before, during, and after the intervention.

DETAILED DESCRIPTION:
Prescreening:

Before the study, the investigators at each site will review existing assessment information for each participant with autism, which may include age, gender, IQ, autism, and behavioral scales, and verbal language functioning to confirm the children that meet the inclusion criteria.

Each dyad's involvement will last over the course of approximately 12 months. The first 3 months will be the intervention and data will be collected throughout. Follow-up data will be collected 3, 6, and 9 months after the intervention is concluded.

The study will involve the following components:

Pre-Assessments：

For children with ASD:

After each dyad is enrolled, the research team assessor/evaluator will administer either the Childhood Autism Rating Scale (CARS) or Autism Diagnostic Observation Schedule (ADOS). Children with ASD in China will be assessed using CARS while the children with ASD will be assessed with ADOS. Further, Vineland Adaptive Behavior Scales will be used for children in both countries

For typically developing children:

The current reading achievement of all typically developing siblings will be assessed by the research team assessor. For siblings in the U.S., DIBELS GK-1 level will be used to assess if the siblings will be able to read words and nonsense words fluently. For siblings in China, different combinations of letters (pinyin) will be assessed.

For parents:

Parents will complete a demographic survey online using their participant ID.

Pretest/Baseline Early literacy: During each session, the research team assessor will ask the children with ASD in the U.S. to read Grade K to Grade 1 letters, words, and nonsense words. If the children could meet the Benchmark goals for core support per DIBELS benchmark goals for Grade K-1, they will then be asked to read a narrative passage for 1 minute and answer questions related to whom, where, and when as well as the actions and internal responses of the characters.

For children with ASD in China, the research team assessor will ask them to read pinyins using the pinyin matrix. If the children could read 70% pinyins correctly, they will then be asked to read a narrative passage with pinyin for 1 minute and answer questions related to whom, where, and when as well as the actions and internal responses of the characters.

Social reciprocity: Parents will place toys, games, and books in a location at home and ask the siblings to play with each other for 15 minutes. The entire 15-minute session will be video recorded and then coded using the Playground Observation of Peer Engagement (POPE) and Reciprocity datasheets.

The assessment for early literacy and social reciprocity skills lasts for a minimum of five days.

Sibling Relationship Quality: Parents will complete one Sibling Inventory of Behavior scale.

Sibling Self-Efficacy scale: The TD sibling will complete a self-efficacy scale.

Sibling and parent interview: The investigators will interview the parents and siblings regarding everyday sibling interaction and relationship and the influence of the sibling with autism on the daily life of the typically developing sibling. The investigators will use some guiding questions to begin the interviews. Questions that elicit additional details or responses for examples and feelings (e.g., Tell me more. How do you feel? Do you have an example?) may be used depending on the answers. The interview will take place online for approximately 1 hour using a teleconference tool (e.g., Zoom), and interviews will be both audio and video recorded.

Random assignments:

In each country, children will be randomly assigned to a treatment-as-usual group and a sibling-mediated intervention group with 10 in each group.

Treatment-as-usual/sibling interaction group:

Parents will place toys, games, and books in a location at home and ask the siblings to spend time with each other for 20-30 minutes, at least three times a week for a total of three months. All sessions will be video recorded. The families in the treatment-as-usual group will receive the intervention after the procedure is completed.

Sibling-mediated intervention group:

The sibling-mediated intervention will start with three 45-minute training sessions for the typically developing sibling via telecommunication (e.g., Zoom) on how to use the model-lead-test strategy (i.e., model the correct response, guided practice of the correct response and test the correct response) and the self-monitoring checklist. During training, parents will be present and may be asked to pretend to be learners.

After the training sessions, the first phase, Compliance Training Phase, will begin. At the beginning of each session, parents will give the TD sibling an activity schedule consisting of the tasks (e.g., a series of questions) for the session. The TD sibling will follow the activity schedule to present the tasks (e.g., asking children with ASD a series of common questions) and use the self-monitoring checklist to deliver model-lead-test when needed. In the initial sessions, the instructor will be present to prompt the TD sibling to deliver the intervention and correctly use the self-monitoring checklist. After each session, the instructor will deliver feedback until the typically developing sibling meets the mastery criterion (i.e., at least 85% correct across five sessions). Once mastery is met, the research team instructor will then review videos every 3-5 days and deliver feedback to the TD sibling. The compliance training phase will last for 9-15 sessions.

During the intervention phase, the research team interventionist will start by briefly meeting with the TD sibling to introduce the self-monitoring checklists for early literacy and social reciprocity. The TD siblings will then follow the visual activity schedule (e.g., the list of the tasks: reading, social play; the order of the activities may change daily) and use the self-monitoring checklists when teaching reading and social reciprocity.

For reading, each week, the investigator will identify 3-5 words in a children's book, the typically developing sibling will read the children's book to the sibling with ASD and pausing upon the target words. The sibling with ASD will be asked to read the target words. If the child with ASD could not read the target words, the typically developing sibling will teach how to read words using model-lead-test. If the child with ASD read the target words correct, the typically developing sibling will provide praise or any other rewards (e.g., high-five, tickle, etc.) as identified by parents. The book will be changed weekly.

For social reciprocity, the parents will bring toys and games and ask the typically developing sibling to play with their sibling with ASD. During the play, after a few physical actions and verbalizations from the typically developing sibling, the typically developing sibling will teach the sibling with ASD to respond with a reciprocal physical action and conversation. If the sibling with ASD responds with a physical action along with conversation, the typically developing sibling will provide praise or any other social rewards.

Similar to the compliance phase, the instructor will initially monitor and deliver feedback over Zoom to the TD sibling in each session until mastery, followed by a variable schedule (e.g., every 3-5 sessions).

Ongoing data collection on the readings and social reciprocity from the children with ASD will be conducted. The compliance training and intervention phases will last 3 months.

Posttest/Post-intervention The procedure for the posttest/post-intervention phase is the same as pretest/baseline phase. In addition, both children in each dyad will complete a social validity questionnaire.

3-month, 6-month, and 9-month follow-ups Three follow-ups will be conducted after 3, 6, and 9 months after the completion of the intervention. The procedure is the same as pretest/baseline phase.

ELIGIBILITY:
Inclusion Criteria:

* Both siblings can demonstrate compliance during instruction.
* Children with ASD can imitate physical actions and repeat vocalizations, answering common questions, label common objects and actions with adjectives.
* Typically developing children can sound out and blend letters during reading.

Exclusion Criteria:

* Children with aggression towards their siblings and noncompliance during instruction
* Children with ASD who can sound out and blend letters.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2025-09-07 (Actual); Study Completion 2025-09-07 (Actual)

PRIMARY OUTCOMES:
Change in oral reading accuracy | Assessment will begin from the date of randomization, during and after the intervention, and up to 9 months after the intervention for a total of approximately 12 months
  Participants in the US will complete DIBELS Grades K-1 Benchmark. Participants in China read pinyin's using a pinyin matrix
Change in social engagement | Assessment will begin from the date of randomization, during and after the intervention, and up to 9 months after the intervention for a total of approximately 12 months
  Children will play with their siblings for 15 minutes. The interaction will be coded using the Playground Observation of Peer Engagement (POPE).
Change in sibling relationship | Assessment will begin from the date of randomization, during and after the intervention, and up to 9 months after the intervention for a total of approximately 12 months
  Parents will complete the "Sibling Inventory of Behavior" scale. The minimum value of the scale is 32, and the maximum value is 160. The scale measures multiple dimensions of the sibling relationship, including companionship, empathy, teaching, rivalry, conflict, avoidance. Higher values obtained in each of the dimensions mean a higher level of companionship, empathy, teaching, rivalry, conflict, or avoidance from the sibling.
Change in sibling self-efficacy. | Assessment will begin from the date of randomization, during and after the intervention, and up to 9 months after the intervention for a total of approximately 12 months
  Typically developing siblings will complete the investigator-created "Children's Self-Efficacy Scale for TD Siblings". The scale is broken down into four sections of four to ten items. Each item is rated from 0 indicating a lack of self-efficacy to 100 indicating confidence. Thus, the minimum score that can be obtained is 0 and the maximum score is 2,700.
Change in reciprocal conversation | Assessment will begin from the date of randomization, during and after the intervention, and up to 9 months after the intervention for a total of approximately 12 months
  Children will play with their siblings for 15 minutes. Components in reciprocal conversation, such as answering questions, expansion, and reciprocal question-asking will be coded.

SECONDARY OUTCOMES:
Change in oral retell | Assessment may begin from the date of randomization, after the intervention, and up to 9 months after the intervention for a total of approximately 12 months
  Participants will read a narrative passage for 1 minute and answer comprehension questions if they pass the DIBELS benchmark or can read pinyin for more than 70% correct
Social validity | Immediately after the intervention
  Both children will complete a social validity survey after the intervention - "Social Validity Survey Questionnaire". The survey is broken into two parts, one for each child in the dyad. All items are rated from 1-5. The minimum score is 14 and the maximum score is 70. However, these items contain positive and negative statements. Thus, a higher (or a lower) score does not necessarily mean a better or worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Chengan Yuan, PhD, Principal Investigator — Arizona State University; Erin Rotheram-Fuller, PhD, Principal Investigator — Arizona State University; Juliet Hart Bartnett, PhD, Principal Investigator — Arizona State University
Locations (3):
- Children's Autism Center, Round Rock, Texas, United States
- China (2):
  - Best Love Child Development Center, Kunming, Yunnan
  - Clover Children Rehabilitation Kindergarten, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Christensen DL, Baio J, Van Naarden Braun K, Bilder D, Charles J, Constantino JN, Daniels J, Durkin MS, Fitzgerald RT, Kurzius-Spencer M, Lee LC, Pettygrove S, Robinson C, Schulz E, Wells C, Wingate MS, Zahorodny W, Yeargin-Allsopp M; Centers for Disease Control and Prevention (CDC). Prevalence and Characteristics of Autism Spectrum Disorder Among Children Aged 8 Years--Autism and Developmental Disabilities Monitoring Network, 11 Sites, United States, 2012. MMWR Surveill Summ. 2016 Apr 1;65(3):1-23. doi: 10.15585/mmwr.ss6503a1. PMID 27031587
- [Background] Johnny L. Matson, Jonathan Wilkins & Jennifer Macken (2008) The Relationship of Challenging Behaviors to Severity and Symptoms of Autism Spectrum Disorders, Journal of Mental Health Research in Intellectual Disabilities, 2:1, 29-44, DOI: 10.1080/19315860802611415
- [Result] Chang YC, Locke J. A systematic review of peer-mediated interventions for children with autism spectrum disorder. Res Autism Spectr Disord. 2016 Jul;27:1-10. doi: 10.1016/j.rasd.2016.03.010. Epub 2016 Mar 26. PMID 27807466
- [Result] Stadnick NA, Stahmer A, Brookman-Frazee L. Preliminary Effectiveness of Project ImPACT: A Parent-Mediated Intervention for Children with Autism Spectrum Disorder Delivered in a Community Program. J Autism Dev Disord. 2015 Jul;45(7):2092-104. doi: 10.1007/s10803-015-2376-y. PMID 25633920
- [Result] Kryzak LA, Jones EA. Sibling self-management: Programming for generalization to improve interactions between typically developing siblings and children with autism spectrum disorders. Dev Neurorehabil. 2017 Nov;20(8):525-537. doi: 10.1080/17518423.2017.1289270. Epub 2017 Mar 9. PMID 28277816
- [Result] Shivers CM, Plavnick JB. Sibling involvement in interventions for individuals with autism spectrum disorders: a systematic review. J Autism Dev Disord. 2015 Mar;45(3):685-96. doi: 10.1007/s10803-014-2222-7. PMID 25178988
- [Result] Archer AL, Hughes CA. Explicit instruction: Effective and efficient teaching. 2011. Guilford Press,